CLINICAL TRIAL: NCT00241514
Title: Efficacy of Esomeprazole 40 mg Once Daily Versus Placebo or Esomeprazole 20 mg Once Daily Versus Placebo in Prevention of Upper Gastrointestinal Symptoms Associated With Continuous Use of NSAIDs Including COX-2 Selective NSAIDs
Brief Title: Esomeprazole for Prevention of Upper Gastrointestinal Symptoms Associated With Continuous Use of NSAIDs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D9617C00002; SH-NEN-0002
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2011-01

CONDITIONS: GERD
Keywords: NSAIDs; Upper GI symptoms
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole

SUMMARY:
This study was a multicentre, double-blind, randomised, placebo-controlled parallel group study consisting of 4 visits over a period of 6 months. The primary variable was to assess the efficacy of esomeprazole 40 mg orally qd (E40) or esomeprazole 20 mg orally qd (E20) versus placebo orally qd after 6 months of treatment for the prevention of relapse of upper GI symptoms associated with NSAID use, including COX-2 selective NSAIDs, in patients receiving daily NSAID therapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Completed the SH-NEN-0001 study with relief of upper GI symptom. Relief is defined as "last 7 days with a diary assessment of None or Minimal, but allowing up to 2 days to be rated as Mild during the 7-day period".
* A clinical diagnosis of a chronic condition (e.g., osteoarthritis or rheumatoid arthritis) that requires continuous daily NSAID treatment for at least 6 months. Daily NSAID treatment is defined as taking the prescribed dose for at least 5 of 7 days in any given week and can include COX-2 selective NSAIDs, multiple NSAIDs, and high-dose NSAIDs.
* Daily NSAID treatment dose and type: (Must have been stable for at least 9 weeks prior to inclusion and; Are expected to remain stable for the duration of the study. and; Must be administered orally. If more than one type of NSAID treatment is used, at least one type must be administered orally).
* Hp negative on Histology performed at baseline endoscopy in the study SHNEN- 0001.

Exclusion Criteria:

* Discontinuation from study SH-NEN-0001
* Pain, discomfort or burning in the upper abdomen precipitated by exercise or relieved by defecation.
* Pain, discomfort or burning in the upper abdomen not associated with the use of NSAIDs, including COX-2 selective NSAIDs.
* Pregnancy or lactation. Women of childbearing potential must maintain effective contraception during the study period as judged by the investigator.
* Need for continuous concomitant therapy with: (Anticoagulants; Corticosteroids at doses higher than explained under inclusion criterion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334
Dates: Start 2001-02; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of esomeprazole 40 mg orally q.d. versus placebo orally q.d.
and 20 mg q.d. versus placebo orally q.d. through 6 months of treatment for the
prevention of relapse of upper GI symptom associated with NSAID use in patients
receiving daily NSAID therapy.

SECONDARY OUTCOMES:
To assess the safety and tolerability of esomeprazole 40 mg orally q.d. versus placebo orally q.d. and 20 mg orally q.d. versus placebo orally q.d. when administered for 6 months to patients receiving daily NSAID therapy.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Nexium Medical Sciences Director, MD, Study Director — AstraZeneca
Locations (113):
- United States (19):
  - Research Site, Tucson, Arizona
  - Research Site, Anaheim, California
  - Research Site, Orange, California
  - Research Site, San Francisco, California
  - Research Site, Bradenton, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, South Miami, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Zephyrhills, Florida
  - Research Site, Conyers, Georgia
  - Research Site, Newburgh, Indiana
  - Research Site, Baltimore, Maryland
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Tulsa, Oklahoma
  - Research Site, Tipton, Pennsylvania
  - Research Site, Norfolk, Virginia
  - Research Site, Virginia Beach, Virginia
- Belgium (29):
  - Research Site, Alleur
  - Research Site, Ans
  - Research Site, Beernem
  - Research Site, Betekom
  - Research Site, Bottelare
  - Research Site, Braine-l'Alleud
  - Research Site, Buizingen
  - Research Site, Duffel
  - Research Site, Durnal
  - Research Site, Erembodegem
  - Research Site, Genk
  - Research Site, Ghent
  - Research Site, Herentals
  - Research Site, Lambermont
  - Research Site, Leut
  - Research Site, Liège
  - Research Site, Linkebeek
  - Research Site, Maasmechelen
  - Research Site, Massemen
  - Research Site, Merelbeke
  - Research Site, Natoye
  - Research Site, Nivelles
  - Research Site, Oud-Heverlee
  - Research Site, Seraing
  - Research Site, Soignies
  - Research Site, Vorst (Brussels)
  - Research Site, Waremme
  - Research Site, Zoersel
  - Research Site, Zolder
- France (19):
  - Research Site, Albens
  - Research Site, Angers
  - Research Site, Dambach-la-Ville
  - Research Site, Dommartin-les-touls
  - Research Site, Fontaine-lès-Dijon
  - Research Site, Gesté
  - Research Site, Gémenos
  - Research Site, Husseren-Wesserling
  - Research Site, La Regrip
  - Research Site, Le Pian-Médoc
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Maromme
  - Research Site, Mont-de-Marsan
  - Research Site, Montingy Les Metz
  - Research Site, Paris
  - Research Site, Saint-Ouen
  - Research Site, Strasbourg
  - Research Site, Tarare
- Germany (27):
  - Research Site, Berlin
  - Research Site, Bernau
  - Research Site, Bochum
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Dresden-Test
  - Research Site, Erfurt
  - Research Site, Erlangen
  - Research Site, Genthin
  - Research Site, Herne
  - Research Site, Kelkheim
  - Research Site, Künzing
  - Research Site, Lienen
  - Research Site, Lüdenscheid
  - Research Site, München
  - Research Site, Münster
  - Research Site, Paderborn
  - Research Site, Passau
  - Research Site, Potsdam
  - Research Site, Ratingen
  - Research Site, Regensburg
  - Research Site, Ribnitz-Damgarten
  - Research Site, Saarbrücken
  - Research Site, Salzgitter
  - Research Site, Wangen
  - Research Site, Wiesbaden
  - Research Site, Wolmirstedt
- Hungary (7):
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Dunaújváros
  - Research Site, Szentes
  - Research Site, Szombathely
  - Research Site, Vác
  - Research Site, Veszprém
- Spain (12):
  - Research Site, Barcelona
  - Research Site, Getafe
  - Research Site, Guadalajara
  - Research Site, Madrid
  - Research Site, Mérida
  - Research Site, Palma de Mallorca
  - Research Site, San Sebastián(Guipuzcoa)
  - Research Site, Seville
  - Research Site, Torrelavega
  - Research Site, Valencia
  - Research Site, Viladecans
  - Research Site, Zaragoza

REFERENCES:
- [Derived] Hawkey CJ, Talley NJ, Scheiman JM, Jones RH, Langstrom G, Naesdal J, Yeomans ND; NASA/SPACE author group. Maintenance treatment with esomeprazole following initial relief of non-steroidal anti-inflammatory drug-associated upper gastrointestinal symptoms: the NASA2 and SPACE2 studies. Arthritis Res Ther. 2007;9(1):R17. doi: 10.1186/ar2124. PMID 17391505